CLINICAL TRIAL: NCT00233753
Title: Cordis Neurovascular Feasibility Study of the Enterprise Self-Expanding Stent System to Facilitate Endovascular Coil Embolization of Wide- Neck Saccular Intracranial Artery Aneurysms
Brief Title: Study of the Enterprise Self-Expanding Stent System With Endovascular Coil Embolization of Wide- Neck Saccular Intracranial Artery Aneurysms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Codman & Shurtleff (Industry)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: USCNVP-01
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2009-01

CONDITIONS: Intracranial, Wide-Neck, Saccular Aneurysms
Keywords: Intracranial; Wide-neck; Saccular; Aneurysms
MeSH Terms: conditions — Aneurysm

INTERVENTIONS:
Device: Cordis Neurovascular Self-Expanding Stent

SUMMARY:
Cordis Self Expanding Stent for use with embolic coils for the treatment of wide-neck, intracranial, saccular aneurysms arising from a parent vessel

ELIGIBILITY:
Inclusion Criteria:

* pts with intracranial, wide-neck, saccular aneurysms

Exclusion Criteria:

* Subject with Hunt and Hess Grade IV or V subarachnoid hemorrhage.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-01; Study Completion 2005-12